CLINICAL TRIAL: NCT05070403
Title: Phase 2 Study of Afatinib in Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Study of Afatinib in Advanced Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20731
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: Skin Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afatinib Intervention (Experimental): Participants will receive afatinib 40 mg once a day. Each cycle is 4 weeks. They will have CT imaging (and/or digital photography) done at baseline and every 8 weeks while on treatment. Participants will have a baseline and on-treatment (at 4 weeks) tumor biopsy, and a biopsy at disease progression if feasible. Patients may remain on treatment as long as they are deriving clinical benefit, until disease progression or intolerable toxicity.
  Interventions: Drug: Afatinib 40 MG

INTERVENTIONS:
Drug: Afatinib 40 MG — Participants will receive 40 mg Afatinib, once daily.

SUMMARY:
The primary purpose of this study is to find out if Afatinib can help treat participants with advanced cSCC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* ECOG performance status ≤2
* Adequate bone marrow, organ function and laboratory parameters:
* ANC ≥ 1.0 × 109/L;
* Hemoglobin ≥ 8 g/dL;
* Platelets ≥ 75 × 109/L;
* AST and ALT ≤5 × ULN
* Calculated creatinine clearance > 15mL/min by Cockroft-Gault formula
* Histologic diagnosis of invasive cutaneous squamous cell carcinoma, that is deemed not appropriate for further surgical intervention and/or radiation therapy. Participants may have either locally advanced or metastatic disease.
* At least 1 measurable lesion - either per RECIST 1.1 criteria, or for patients with externally visible cuSCC lesion(s) not measurable on imaging, at least one lesion ≥1 cm in longer diameter, amenable to digital photography with bi-dimensional measurements
* Participants must have received prior immunotherapy with an anti-PD-1/PD-L1 antibody, if participant was deemed eligible (i.e., was not immunosuppressed or a transplant receipt, etc)
* Immunosuppressed participant including those with concurrent autoimmune diseases and solid organ transplant recipients are eligible
* Prior to first dose of study treatment, participant must be at least 2 weeks from any prior systemic therapy, major surgery or radiation
* Able to undergo a pre-treatment and on-treatment tumor biopsy
* Female participants of childbearing potential must have a negative serum or urine β-HCG test result. Female participants of childbearing potential and male participants must agree to use methods of contraception that are highly effective.
* Participants with brain metastases are permitted assuming that the brain metastases have been adequately treated with prior surgery or radiation.

Exclusion Criteria:

* In participants with known liver cirrhosis, those with severe (Child Pugh C) hepatic impairment will be excluded.
* Untreated, uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable or require corticosteroids,
* Participants with mixed histologies (eg, sarcomatoid, adenosquamous) will generally not be eligible, unless the predominant histology is invasive cuSCC.
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to randomization. Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load prior to randomization.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 1 Year
  Overall response rate (ORR) as defined by proportion of patients who have achieved a complete or partial response per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival | Up to 5 Years
  Progression free survival, defined as the time from first dose to the earlier date of assessment of progression or death by any cause in the absence of progression
Overall survival | Up to 5 Years
  Overall survival, as measured from the date of first dose to the date of death by any cause
Treatment-related adverse events | Up to 40 days after end of treatment
  Treatment-related adverse events per NCI CTCAE v5 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=20731